CLINICAL TRIAL: NCT06259721
Title: Efficacy and Safety of Anti-PD1 Monoclonal Antibody Combined With Nimotuzumab and Capecitabine in Patients With First-line Platinum-resistant Recurrent/Metastatic Nasopharyngeal Carcinoma: A Single-arm, Open-label, Multi-center Phase II Clinical Trial
Brief Title: Anti-PD1 Monoclonal Antibody Combined With Nimotuzumab and Capecitabine in Patients With First-line Platinum-resistant Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INC-RMNPC
Record Dates: First submitted 2024-02-07; First posted 2024-02-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; anti-PD1 antibody; Nimotuzumab; Capecitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination Treatment (Experimental)
  Interventions: Drug: Anti-PD1 antibody, nimotuzumab and capecitabine

INTERVENTIONS:
Drug: Anti-PD1 antibody, nimotuzumab and capecitabine — Combination phase Anti-PD1 monoclonal antibody: Choose one of the anti-PD-1 monoclonal antibody drugs reimbursed by medical insurance, toripalimab (240mg), camrelizumab (200mg), tislelizumab (200mg) or others; Intravenous infusion, every 3 weeks .
  Nimotuzumab:: In the first 6 cycles, 200 mg, intravenous infusion, every 1 week, and 400 mg is administered for the first time.
  Capecitabine: 1000 mg/m2, orally twice daily on days 1-14, every 3 weeks
  Maintenance phase:
  Anti-PD1 monoclonal antibody: anti-PD-1 monoclonal antibody drugs, Intravenous infusion, every 3 weeks.
  Nimotuzumab treatment: 400 mg, intravenous infusion, every 3 weeks. Capecitabine: 1000 mg/m2, orally twice daily on days 1-14, every 3 weeks；
  The duration of treatment is 1 year or until intolerable toxic reactions occur, or disease progresses, or the patient withdraws consent, or the investigator determines that the patient needs to withdraw from treatment.

SUMMARY:
The purpose of this study is to explore the efficacy and safety of a combination regimen of Anti-PD1 monoclonal antibody, nimotuzumab, and capecitabin in treating recurrent or metastatic nasopharyngeal carcinoma patients who have failed first-line platinum-based chemotherapy.

DETAILED DESCRIPTION:
Currently, there is still no uniform treatment regimen for treating recurrent or metastatic nasopharyngeal carcinoma patients who failed to first-line platinum-based chemotherapy. Anti-PD-1 monoclonal antibody showed efficacy and safety in previous studies, however, the efficacy of immunotherapy alone was limited. Immunotherapy combined with other treatment regimens for recurrent or metastatic nasopharyngeal carcinoma is a strategy that needs to be urgently explored. Epidermal growth factor receptor (EGFR) is an important target in the treatment of nasopharyngeal carcinoma. Nimotuzumab, an EGRF antibody selectively inhibits epidermal growth factor receptors, has shown strong clinical utility in Nasopharyngeal Carcinoma. Nimotuzumab is an IgG1 monoclonal antibody targeting EGFR. It can not only effectively block the EGFR signaling pathway to promote cell death, but also activate immunity through ADCC to mediate anti-tumor effects.

Anti-PD-1 antibodies relieve inhibition of cytotoxic lymphocytes to promote tumor regression. Nimotuzumab targeting EGFR mediates antibody-dependent cellular cytotoxicity and promotes communication between immune cells, including natural killer and dendritic cells. This communication can trigger tumor antigen-specific cellular immunity and generate antigen-specific T lymphocyte responses. Furthermore, therefore, recruitment of adaptive and innate immunity and antibody-dependent cellular cytotoxicity may induce antitumor synergy. Considering that anti-PD1 monoclonal antibodies and nimotuzumab play a synergistic role in enhancing anti-tumor immunity. The combination of anti-EGFR monoclonal antibody and anti-PD-1 monoclonal antibody has shown good efficacy in recurrent and metastatic head and neck squamous cell carcinoma. The overall response rate (ORR) of the combination treatment reached 45%, better than the ORR of the anti-PD-1 monoclonal antibody alone (20%).

As a new type of fluorouracil oral anticancer drug, capecitabine has better efficacy and lower toxicity than 5-Fu [14]. Two recent clinical trials have confirmed that maintenance therapy with capecitabine oral chemotherapy can effectively reduce the risk of metastasis in locally advanced nasopharyngeal carcinoma, suggesting that new fluorouracil drugs have good anti-cancer effects. Clinical studies from recurrent metastatic nasopharyngeal carcinoma also confirmed that capecitabine metronomic therapy can improve overall survival. Maintenance chemotherapy is a strategy of administering cytotoxic drugs at high frequency, low doses, and minimal downtime.

Based on this, this study aims to evaluate the efficacy and safety of anti-PD1 monoclonal antibody combined with nimotuzumab and capecitabine in patients with recurrent or metastatic nasopharyngeal carcinoma who failed to first-line platinum-based chemotherapy, to provide new evidence for individualized comprehensive treatment in nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed with recurrent or metastatic nasopharyngeal carcinoma which is not amenable to curative treatment with surgery and/or radiation therapy. If the patient refuses biopsy of metastatic lesions, those diagnosed with metastasis based on imaging evidence and clinical evidence can be enrolled.
2. Have failed for first-line platinum-based chemotherapy. Previously received first-line platinum-based chemotherapy for recurrent or metastatic disease and had disease progression during or after treatment; or recurrence and metastases within 6 months after treatment of platinum-based chemoradiation.
3. Age ≥ 18 years and ≤ 75 years, both genders.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
5. The life expectancy of at least 3 months.
6. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria.
7. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment) as determined by:

   Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L; Hemoglobin ≥ 9 g/dL; serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN), (for subjects with liver metastases, TBIL ≤3×ULN; ALT and AST≤5×ULN); Creatinine ≤1.5×ULN or creatinine clearance rate≥50 ml/min (Cockcroft-Gault formula); serum albumin ≥28 g/L; Thyroid-stimulating hormone (TSH) levels ≤1×ULN (however, patients with free Triiodothyronine [FT3] or free Thyroxine [FT4] levels ≤1× ULN may be enrolled); INR, APTT≤1.5 x ULN.
8. All women with fertility potential must undergo a urine or serum pregnancy test during screening and the results are negative.
9. Written informed consent.

Exclusion Criteria:

* 1. Those with a history of severe immediate allergy to any drugs used in this study; 2. Patients who have previously received anti-EGFR monoclonal antibodies (nitolizumab, cetuximab) and anti-PD-1 monoclonal antibodies.

  3. Combined with other malignant tumors; 4. Any of the following conditions exist within 6 months before screening: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident, transient cerebral ischemia Paroxysmal or symptomatic pulmonary embolism. Patients with known coronary artery disease, congestive heart failure that does not meet the above criteria, or left ventricular ejection fraction <50% must be treated with an optimized and stable medical regimen as determined by the treating physician, who may consult a cardiologist if appropriate; 5. Patients who have received any of the following treatments:

  (1) Have received any investigational drugs within 4 weeks before using the investigational drugs for the first time; (2) Use of large amounts of glucocorticoids or other immunosuppressants (including but not limited to prednisone, dexamethasone, azathioprine, methotrexate, thalidomide and anti-tumor necrosis factor within 4 weeks before treatment (drugs against TNF), or subjects who require hormonal therapy during clinical trials. Other special circumstances need to be communicated with the sponsor. In the absence of active autoimmune disease, inhaled or topical steroids and adrenocortical hormone replacement at doses >10 mg/day prednisone therapeutic dose are allowed; (4) Those who have received anti-tumor vaccines or have received live vaccines within 4 weeks before the first administration of the study drug; (5) Have undergone major surgery or serious trauma within 4 weeks before using the study drug for the first time; (6) Enroll in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up; 6. Patients with active autoimmune diseases or a history of autoimmune diseases that may relapse

Note: Patients with the following diseases are not excluded and can enter further screening:

1. Controlled type 1 diabetes
2. Hypothyroidism (if it can be controlled with hormone replacement therapy alone)
3. Skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, alopecia)
4. Any other disease that is not expected to recur in the absence of external triggers 7. Active infections, including tuberculosis, hepatitis B, hepatitis C and human immunodeficiency virus. Patients with positive HBV surface antigen (HBsAg) but HBV DNA <1000 copies/mL are eligible to participate in this study; patients with positive HCV antibody test results can only participate if the HCV RNA polymerase chain reaction test result is negative. Selected for this study; 8. History of idiopathic pulmonary fibrosis, drug-induced pneumonia, organizing pneumonia (bronchiolitis obliterans), idiopathic pneumonia or evidence of active pneumonia on chest CT scan during screening; 9. No capacity for civil conduct or limited capacity for civil conduct; 10. Drug abuse or alcohol addiction, the patient has physical or mental illness, and the researcher believes that the patient cannot fully or fully understand the possible complications of this study; 11. Other serious acute or chronic medical conditions that may increase the risks related to the treatment of the research protocol, or may interfere with the interpretation of the research results and (according to the investigator's judgment) may make the patient unfit to participate in this study (including immune colitis, inflammatory colitis, Enteropathy, non-infectious pneumonia, pulmonary fibrosis) or mental illness (including dementia and epilepsy, suicidal ideation or behavior recently, within the past year, or active) or abnormal laboratory tests; 12. Previously diagnosed with immunodeficiency or known diseases related to human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS); 13. Pregnant or lactating female patients, male or female patients with childbearing potential but unwilling or unable to use contraception during the entire study period and for at least 1 year after the end of the treatment plan; 14. Those with recurrent nasopharyngeal carcinoma are suitable for surgical treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-08-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 months
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI) An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI) An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI)

SECONDARY OUTCOMES:
Disease control rate | 6 months
  A disease control rate is defined as either a confirmed CR or a PR or a SD, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI).
Duration of response | 1 year
  Defined from date of first confirmed CR or a PR to date of first documentation of progression or death due to any cause, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute
Overall survival rate | 2 years
  Defined from date of registration to date of first documentation of death from any cause oDefined from date of registration to date of first documentation of death from any cause or censored at the date of the last follow-up.
  r censored at the date of the last follow-up.
Progression-free survival rate | 2 years
  Defined from date of registration to date of first documentation of progression or death due to any cause.
Incidence rate of adverse events (AEs) | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jingao Li, MD, Principal Investigator — NHC Key Laboratory of Personalized Diagnosis and Treatment of Nasopharyngeal Carcinoma, Jiangxi Cancer Hospital
Locations (1):
- Department of Nasopharyngeal Carcinoma, Jiangxi Cancer Hospital, Nanchang, Jiangxi, China